CLINICAL TRIAL: NCT03276780
Title: NRT Sampling and Selection to Increase Medication Adherence
Brief Title: Nicotine Replacement Therapy (NRT) Sampling and Selection to Increase Medication Adherence
Acronym: NRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Karen Cropsey, Professor of Psychiatry, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F151019004; R34DA043346 (NIH)
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Results first posted 2021-12-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: In vivo or standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- In vivo (Experimental): Will receive 4 types of short-acting NRT medication to use in combination with the nicotine patch in each counseling session for four sessions. At the fifth session, participants will select their short acting NRT to use with the patch to make a cessation attempt.
  Interventions: Behavioral: Counseling; Drug: combination NRT
- Standard of care (Active Comparator): Will receive 4 sessions of behavioral counseling around their smoking. At the fifth session, participants will select their short-acting NRT to use with the nicotine patch based on a product description of each product to make a cessation attempt.
  Interventions: Behavioral: Counseling; Drug: combination NRT

INTERVENTIONS:
Behavioral: Counseling — Both groups receive smoking cessation counseling although one is focused on medication adherence and addressing barriers to adherence while the other is focused on standard behavioral strategies to quit smoking
Drug: combination NRT — Both groups will receive combination NRT to help with smoking cessation

SUMMARY:
To determine the preliminary impact on Nicotine Replacement Therapy (NRT)adherence and examine the underlying mechanisms of action associated with adherence.

DETAILED DESCRIPTION:
Adherence is a critical target for successful smoking cessation, with good adherence associated with a three-fold increase in cessation rates relative to poor adherence. Psychoeducational interventions focused on increasing adherence to NRT do not result in behavioral change (e.g., smoking cessation). Experiential approaches, such NRT sampling with practice quit attempts (PQAs), are based on learning theory models of behavioral change and have resulted in increased motivation, self-efficacy, adherence, and abstinence relative to psychoeducation or motivational interventions. However, nicotine sampling still relies of the participant using NRT outside of session, which may not occur. Providing an experiential intervention in which the NRT is sampled and any problems with NRT reframed during the session may provide a powerful learning experience that can increase in home sampling with PQAs and long-term adherence, ultimately increasing the likelihood of smoking cessation. This may be particularly relevant for low-income smokers who hold more negative views of NRT, have lower health literacy, and are less likely to use medication during cessation attempts.

ELIGIBILITY:
Inclusion Criteria:

a) 18 years or older; b) qualifying as low income (as defined by making <150% above the poverty line or <$22,260 as a single or <$45,570 for a family of four); c) Smoking at least 5 cigarettes per day (CPD) for the past year and a carbon monoxide (CO) level of less than 8 ppm to ensure daily smoking. This relatively low cutoff was chosen due to the expectation of enrolling a large >50% African-American who average <10 CPD compared to Whites who average ~15 CPD.; and d) English speaking.

Exclusion Criteria:

a) Living in a restricted environment (e.g., prison or jail facility, etc.); b) Pregnant or nursing (all women will be required to use an acceptable form of contraception); c) Currently enrolled in a smoking cessation treatment program, using NRT products, or prescribed bupropion or varenicline; d) Known allergy to any of the nicotine replacement products or sensitivity to adhesive used in nicotine patches; e) Trouble breathing, a pulmonary condition, or sinus problems; f) Within one month post-myocardial infarction or untreated severe angina; g) poor dentation or temporomandibular joint (TMJ) problems such as unable to use nicotine gum; h) Cognitive impairment or unstable psychiatric condition that interferes with the informed consent process (individuals stable on psychiatric medications will be included); or i) Daily or exclusive use of other tobacco products (e.g., electronic cigarettes, little cigars, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cropsey, PsyD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sisson ML, Gajos JM, Wolford-Clevenger C, Chichester KR, Hawes ES, Hill SV, Shelton RC, Hendricks PS, Businelle MS, Carpenter MJ, Cropsey KL. Impact of Nicotine Replacement Therapy Sampling on Cessation-Related Processes. J Addict Med. 2024 Jul-Aug 01;18(4):397-403. doi: 10.1097/ADM.0000000000001298. Epub 2024 Mar 6. PMID 38446860

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | In Vivo | Standard of Care
Started | 41 | 39
Completed | 23 | 29
Not Completed | 18 | 10
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 3 | 5
Not completed — Moved out of state | 1 | 1
Not completed — Already enrolled in another smoking cessation study providing NRT | 1 | 0
Not completed — No show to appointments after baseline through Week 5 | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In Vivo | Standard of Care | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Categorical [Count of Participants; unit: Participants] — Demographic information was collected using the Demographic Form, a measure developed in the research lab (i.e. no standardized scoring). This measure was used to collect demographic information about the participant, including age, sex, ethnicity, and race.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 41 | 39 | 80
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic information was collected using the Demographic Form, a measure developed in the research lab (i.e. no standardized scoring). This measure was used to collect demographic information about the participant, including age, sex, ethnicity, and race.
  Participants
    Female | 18 | 12 | 30
    Male | 23 | 27 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Demographic information was collected using the Demographic Form, a measure developed in the research lab (i.e. no standardized scoring). This measure was used to collect demographic information about the participant, including age, sex, ethnicity, and race.
  Participants
    Hispanic or Latino | 2 | 0 | 2
    Not Hispanic or Latino | 39 | 39 | 78
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Demographic information was collected using the Demographic Form, a measure developed in the research lab (i.e. no standardized scoring). This measure was used to collect demographic information about the participant, including age, sex, ethnicity, and race.
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 22 | 23 | 45
    White | 18 | 15 | 33
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 39 | 80
Quitting Smoking Behaviors at Baseline [Count of Participants; unit: Participants] — Quitting smoking behaviors was measured using the Smoking History Form, a measure developed in the research lab (i.e. no standardized scoring). This measure was used as a demographic form to collect information about participant history of smoking behaviors and quitting smoking behaviors.
  Participants
    Thinking of quitting smoking in the next month | 24 | 21 | 45
    Thinking of quitting smoking within the next 6 months | 17 | 14 | 31
    Tried NRT to help quit smoking before? | 13 | 16 | 29
    Tried therapy to help quit smoking before? | 2 | 1 | 3
    Tried self-help materials to help quit before? | 1 | 4 | 5
    Tried hypnosis to help quit smoking before? | 2 | 0 | 2
    Tried medication to help quit smoking before? | 4 | 7 | 11
    Tried e-cigarettes to help quit smoking before? | 12 | 12 | 24
    Are any medical problems worsened by smoking? | 4 | 10 | 14
    Live with people who smoke? | 29 | 29 | 58
    Not thinking of quitting smoking | 0 | 4 | 4
Cigarettes Per Day at Baseline [Mean (Standard Deviation); unit: cigarettes per day] | 19.46 (11.05) | 18.36 (9.26) | 18.93 (10.17)
Carbon Monoxide (CO) Level at Baseline [Mean (Standard Deviation); unit: parts per million (ppm) of CO] | 18.56 (11.28) | 18.23 (8.02) | 18.40 (9.76)
Number of Years Smoked Reported at Baseline [Mean (Standard Deviation); unit: years] | 24.73 (11.18) | 28.92 (10.82) | 26.79 (11.13)
Intensity of Nicotine Dependency at Baseline [Mean (Standard Deviation); unit: scores on a scale] — Fagerstrom Test for Nicotine Dependence (FTND) is a standardized instrument for assessing the intensity of physical addiction to nicotine. The FTND contains six items containing yes/no items and multiple choice items. Yes/no items are scored from 0 to 1, and the multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0 to 10. The lowest score on the FTND is a 0, and the highest score on the FTND is a 10. The higher the total FTND score, the worse the participants' outcome is since this indicates a greater intensity of physical dependency on nicotine.
  scores on a scale | 6.49 (1.79) | 6.0 (1.84) | 6.26 (1.79)
Smoking Urges at Baseline [Mean (Standard Deviation); unit: units on a scale] — Participant smoking urges were assessed using the Questionnaire of Smoking Urges (QSU), which is a standardized assessment used to determine level of cravings for smoking. There are ten items in this assessment, and each item was rated on a scale from 1 (strongly disagree) to 7 (strongly agree). The items are summed to determine a total score for level of smoking urges. The lowest score on this scale is 10, and the highest score on the scale is 70. Higher scores indicate worse outcomes for the participant since higher scores indicate more intense smoking urges.
  units on a scale | 46.07 (15.54) | 44.36 (16.58) | 45.24 (15.98)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Participant Retention
Description: Feasibility of the novel NRT intervention was measured by enrolling the targeted sample size of 80 participants. This outcome measure was also measured by the rate of retention of the participants from baseline to the last study visit after 4 months had passed.
Time Frame: From baseline through 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 41 | 39
Participants
  Participant retention rate | 23 | 29
  Participant attrition rate | 18 | 10

2. Primary Outcome: Rate of Recruitment
Description: The acceptability of the novel NRT intervention was measured by calculating the rate of recruitment of study participants during the 56 weeks of active recruitment and intervention for this study.
Time Frame: 56 weeks
Measure: Number; unit: participants screened per week
Groups:
- Total Participants Screened: The total number of participants who were screened for potential enrollment in the study.
Arm/Group | Total Participants Screened
Number analyzed (Participants) | 327
participants screened per week | 5.84

3. Primary Outcome: Rate of Enrollment
Description: The acceptability of the novel NRT intervention was measured by calculating the rate of enrollment of study participants during the 56 weeks of active recruitment and intervention for this study.
Time Frame: 56 weeks
Measure: Number; unit: participants enrolled per week
Groups:
- Total Participants Enrolled: The total number of participants enrolled in the study.
Arm/Group | Total Participants Enrolled
Number analyzed (Participants) | 80
participants enrolled per week | 1.43

4. Primary Outcome: Treatment Satisfaction
Description: Treatment satisfaction was measured using the Treatment Satisfaction Survey (TSS), a measure developed in the research lab (i.e. no standardized scoring). The measure included 10 questions about satisfaction with the study treatment that participants rated from 1 (not helpful) to 7 (very helpful). The minimum value for this scale was 10 and the maximum value for this scale was 70, with a total score of 70 indicating greater satisfaction with the study treatment and a score of 10 indicating no satisfaction with the study treatment. Higher scores on this measure indicated better outcomes for the participant since higher scores indicated more satisfaction with the study treatment.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 27 | 35
score on a scale | 67.70 (3.81) | 69.20 (4.81)

5. Primary Outcome: Treatment Satisfaction
Description: as for outcome 4
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 23 | 31
score on a scale | 65.21 (10.67) | 66.39 (5.91)

6. Primary Outcome: Treatment Satisfaction
Description: as for outcome 4
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 29 | 23
score on a scale | 66.35 (9.82) | 65.62 (10.57)

7. Primary Outcome: Treatment Expectancies at Baseline
Description: Treatment expectancies were measured using the Treatment Expectations questionnaire, a measure developed in the research lab (i.e. no standardized scoring). This measure included 8 items assessing how useful participants' believed the study treatment would be in helping them quit smoking. Participants rated items 1-5 on a scale from 1 (not at all helpful) to 7 (very much helpful). For items 1-3, participants chose which study treatment they would recommend the most to a friend (i.e. the nicotine patch, nicotine gum, nicotine inhaler, nicotine nasal spray, nicotine lozenge, or none), which study treatment they would recommend least to a friend, and overall, which study treatment they found to be the most useful. Only items 1-5 were analyzed for outcomes, with 35 as the maximum value and 5 as the minimum value. Higher scores indicated higher participant expectations for the study treatment and higher expectations for their treatment outcome.
Time Frame: Assessed at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 21 | 22
score on a scale | 23.29 (7.68) | 21.23 (10.58)

8. Primary Outcome: Treatment Credibility
Description: Treatment credibility was measured using the Credibility and Expectancy Questionnaire (CEQ), which is a standardized measure of treatment credibility and expectancy. CEQ scores were standardized, with the minimum score being -13.5 and the maximum score being 4.43. Higher scores indicated the participant believed the treatment was more credible and had higher expectations for their treatment outcome.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 27 | 35
score on a scale | 1.43 (3.67) | 0.84 (5.05)

9. Primary Outcome: Treatment Credibility
Description: Treatment credibility was measured using the Credibility and Expectancy Questionnaire (CEQ), which is a standardized measure of treatment credibility and expectancy. CEQ scores were standardized, with the minimum score being -13.5 and the maximum score being 4.43. High scores indicated the participant believed the treatment was more credible and had higher expectations for their treatment outcome.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 23 | 31
score on a scale | -0.74 (5.12) | 0.08 (3.78)

10. Primary Outcome: Treatment Credibility
Description: as for outcome 9
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 23 | 29
score on scale | -0.26 (5.22) | -1.64 (5.47)

11. Primary Outcome: Number of Participants With Medication Adherence at Week 6
Description: Medication adherence was assessed through self reports from participants and confirmed with package counts by study staff.
Time Frame: From baseline through 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 26 | 34
Participants
  No patch doses missed | 22 | 26
  No NRT doses missed | 23 | 27

12. Primary Outcome: Number of Participants With Medication Adherence at Week 9
Description: as for outcome 11
Time Frame: From baseline through 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 26 | 33
Participants
  No patch doses missed | 23 | 24
  No NRT doses missed | 26 | 33

13. Primary Outcome: Number of Participants With Medication Adherence at Week 13
Description: as for outcome 11
Time Frame: From baseline through 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | In Vivo | Standard of Care
Number analyzed (Participants) | 21 | 30
Participants
  No patch doses missed | 18 | 21
  No NRT doses missed | 17 | 22

ADVERSE EVENTS:
Time Frame: Baseline through 4 months
Arm/Group | In Vivo | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/39
Other Adverse Events (participants affected / at risk) | 15/41 | 2/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In Vivo (N=41) | Standard of Care (N=39)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Participant was hospitalized for treatment for pneumonia between baseline and the first intervention session. Participant was unable to complete the first intervention session for 3 weeks.
Severe Depression (Psychiatric disorders) | 0 (0) | 1 (1) — Participant was admitted to inpatient psychiatric treatment for symptoms of depression between baseline and the first intervention session. Participant was unable to complete the first intervention session for 3 weeks.
Undisclosed Virus (General disorders) | 1 (1) | 0 (0) — Participant reported being hospitalized to be treated for an undisclosed virus between sessions.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In Vivo (N=41) | Standard of Care (N=39)
Nasal Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Occurred while using the nicotine nasal spray.
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Occurred while using the nicotine nasal spray.
Nasal Drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Occurred while using the nicotine nasal spray.
Ear Pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) — Occurred while using the nicotine nasal spray. 1 instance occurred without any NRT use (not related to study medication).
Excessive Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Occurred while using the nicotine nasal spray.
Nicotine Dosage Too Strong (General disorders) | 1 (1) | 0 (0) — Occurred while using the nicotine gum.
Vivid Dreams/Nightmares (General disorders) | 4 (4) | 0 (0) — Occurred while using either the 21 mg patch or 14 mg patch.
Burning Mouth/Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Occurred while using the 2 mg or 4 mg nicotine lozenges/gum or the nicotine inhaler
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — Occurred while using the 21 mg or 14 mg nicotine patch. 1 participant reported an unrelated neck rash while using the 4 mg and 2 mg nicotine lozenges.
Excessive Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Occurred when using the nicotine inhaler.
Headache (General disorders) | 2 (2) | 1 (1) — Occurred when using the nicotine patches and nicotine lozenges in combination, as well as when using the nicotine inhaler.
Stomach ache (Gastrointestinal disorders) | 0 (0) | 1 (1) — Occurred when using the nicotine patches and nicotine lozenges in combination.
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) — Occurred after using the nicotine patch, nicotine inhaler, nicotine gum, and nicotine lozenges.
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) — Occurred when using the nicotine replacement products.
Nasal Burning (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Occurred when using the nicotine nasal spray.
Nasal Tingling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Occurred when using the nicotine nasal spray.
Jitteriness (General disorders) | 1 (1) | 0 (0) — Occurred when using the nicotine inhaler.
Nasal Blistering (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Occurred when using the nicotine nasal spray.
Watering Eyes (Eye disorders) | 1 (1) | 0 (0) — Occurred when using the nicotine nasal spray.
Increased Heart Rate (General disorders) | 1 (1) | 0 (0) — Occurred when using the nicotine nasal spray.
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — A participant reported being treated for an upper respiratory infection. This infection was unrelated to the participant using any study NRT medication.
Tooth Pain (General disorders) | 1 (1) | 0 (0) — Participant reported tooth pain during session that was not related to using the study NRT medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT03276780/Prot_001.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT03276780/SAP_002.pdf